| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
|---|---|
| Detailed Title: | A Phase IIIB, non-randomized, open-label, multi-country, multi-centric cross-vaccination study to evaluate the safety of GSK Biologicals' Herpes Zoster subunit (HZ/su) vaccine when administered intramuscularly on a two-dose schedule to subjects who previously received placebo in ZOSTER-006 and ZOSTER-022 studies. |
| eTrack study number and<br>Abbreviated Title | 204486 (ZOSTER-056) |
| Scope: | All data pertaining to the above study. |
| Date of Statistical Analysis<br>Plan | Final: 26-Feb-2019 |
| Co-ordinating author: | (Expert Biostatistician), PPD (Expert Statistician) |
| Reviewed by: | Clinical and Epidemiology Project Lead) PPD (Clinical Research and Development Lead) PPD (Clinical Research and Development Lead) PPD (Lead statistician) PPD (Lead statistical analyst) PPD (Scientific writer) PPD (Regulatory Affairs) PPD (SERM Scientist) PPD (Public disclosure representative) |
| Approved by: | Clinical and Epidemiology Project Lead) PPD (Clinical Research and Development Lead) PPD (Lead statistician) PPD (Lead statistical analyst) (Scientific writer) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 14 April 2017)

204486 (ZOSTER-056) Statistical Analysis Plan Final

#### **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| LIS | ST OF ABBREVIATIONS | | 9 |
| 1. | DOCUMENT HISTORY | | 10 |
| 2. | STUDY DESIGN | | 10 |
| 3. | OR IECTIVES | | 12 |
| ٥. | | | |
| 4. | ENDPOINTS | | 12 |
| 5. | ANALYSIS SETS | | 13 |
| | | d Cohort | |
| | 5.2. Criteria for eliminating da | ta from Analysis Sets | 13 |
| | | n Total Vaccinated Cohort (TVC)uded subjects | |
| _ | | • | |
| 6. | | | |
| | 6.1.1. Analysis of dem | nographics/baseline characteristics planned | |
| | | iderations | |
| | - <b>I</b> | ocure planned in the protocol | |
| | | osure planned in the protocoliderations | |
| | | idel allol 15 | |
| | | ety planned in the protocol | |
| | | iderations | |
| | | 'incidence | |
| | | pected HZ incidence planned in Protocol | |
| | 6.4.2. Additional cons | ideration | 17 |
| 7. | ANALYSIS INTERPRETATION | | 17 |
| 8. | CONDLICT OF ANALYSES | | 17 |
| Ο. | | | |
| | | for interim analyses | |
| 9. | CHANGES FROM PLANNED AN | NALYSES | 17 |
| 10. | ). LIST OF FINAL REPORT TABLE | ES, LISTINGS AND FIGURES | 18 |
| 11. | . ANNEX 1 STANDARD DATA DE | ERIVATION RULES AND STATISTICAL | |
| | METHODS | | |
| | 11.1. Statistical Method Refere | nces | 19 |

| | | | | 204486 (ZOSTER-056)<br>Statistical Analysis Plan Final |
|---|---|---|---|---|
| | 11.2. | | d data derivation<br>Date derivation | 19 |
| | | | Dose number Demography | |
| | 11.3. | 11.2.4. | Safetyof Decimals | 20 |
| 12. | ANNE | X 2: SUM | MARY ON ELIMINATION CODES | 21 |
| | | | DY SPECIFIC MOCK TFLe of Tables and Figures | |

204486 (ZOSTER-056) Statistical Analysis Plan Final

#### **LIST OF TABLES**

| | | PAGE |
|---------|--------------------------------------------------|------|
| Table 1 | Study groups and epochs foreseen in the study | 10 |
| Table 2 | Study groups and treatment foreseen in the study | 11 |
| Table 3 | Blinding of study epochs | 11 |

204486 (ZOSTER-056) Statistical Analysis Plan Final

#### LIST OF TEMPLATES

| | | PAGE |
|---|---|---|
| Template 1 | Study population (Total Vaccinated Cohort) | 21 |
| Template 2 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Total Vaccinated Cohort) | 22 |
| Template 3 | Summary of demographic characteristics (Total Vaccinated Cohort) | 22 |
| Template 4 | Number of subjects by center (Total Vaccinated Cohort) | 23 |
| Template 5 | Number of subjects enrolled into the study as well as the number excluded from TVC analysis with reasons for exclusion | 23 |
| Template 6 | Number of subjects at each visit and list of withdrawn subjects (Total Vaccinated Cohort) | 23 |
| Template 7 | List of subjects withdrawn from vaccination with reason for withdrawal (Total Vaccinated Cohort) | 23 |
| Template 8 | Deviations from specifications for intervals between study visits (Total Vaccinated Cohort) | 24 |
| Template 9 | Number of enrolled subjects by country | 24 |
| Template 10 | Number of enrolled subjects by age category | 24 |
| Template 11 | Minimum and maximum activity dates (Total Vaccinated Cohort) | 24 |
| Template 12 | Study population – by age sub-group (Total Vaccinated Cohort) | 25 |
| Template 13 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal – by age sub-group (Total Vaccinated Cohort) | 25 |
| Template 14 | Summary of demographic characteristics - by age sub-group (Total Vaccinated Cohort) | 26 |
| Template 15 | Number of subjects by center - by age sub-group (Total Vaccinated Cohort) | 26 |
| Template 16 | Number of subjects at each visit and list of withdrawn subjects by - age sub-group (Total Vaccinated Cohort) | 27 |
| Template 17 | Number and percentage of subjects who received study vaccine doses (Total Vaccinated Cohort) | 27 |
| Template 18 | Number and percentage of subjects reporting the occurrence of<br><grade 3=""> <non-serious><unsolicited adverse="" events=""> classified<br/>by MedDRA Primary System Organ Class and Preferred Term</unsolicited></non-serious></grade> | |

204486 (ZOSTER-056) Statistical Analysis Plan Final

| | <with causal="" relationship="" to="" vaccination=""> <with attended="" medically="" visit=""> within the 30-day (Days 0-29) post-vaccination period (<total -="" 022="" cohort="" cohort,="" confirmed="" during="" episode="" hz="" total="" vaccinated="" zoster-006="">)</total></with></with> | 27 |
|---|---|---|
| Template 19 | Number and percentage of doses with <grade 3=""> unsolicited adverse events classified by MedDRA Primary System Organ Class and Preferred Term <with causal="" relationship="" to="" vaccination=""> <with attended="" medically="" visit=""> within the 30-day (Days 0-29) post-vaccination period (Total Vaccinated Cohort)</with></with></grade> | 28 |
| Template 20 | Global summary of <grade 3=""> <non-serious><unsolicited adverse="" events=""> <with causal="" relationship="" to="" vaccination=""> <with attended="" medically="" visit=""> reported within the 30-day (Days 0-29) post-vaccination period (Total Vaccinated Cohort)</with></with></unsolicited></non-serious></grade> | 28 |
| Template 21 | Number and percentage of subjects reporting the occurrence of <potential diseases="" immune-mediated=""> <serious adverse="" events=""> classified by MedDRA Primary System Organ Class and Preferred Term <with causal="" relationship="" to="" vaccination=""> reported <from 30="" days="" dose="" first="" last="" post="" to="" up="" vaccination=""> <after 30="" days="" dose="" end="" last="" post="" study="" to="" up="" vaccination=""> <from end="" first="" study="" until="" vaccination=""> (<total -="" 022="" cohort="" cohort,="" confirmed="" during="" episode="" hz="" total="" vaccinated="" zoster-006="">)</total></from></after></from></with></serious></potential> | 29 |
| Template 22 | Number and percentage of subjects <with><experiencing> fatal SAEs classified by MedDRA Primary System Organ Class and Preferred Term <who died=""> <with fatal="" of="" onset="" sae=""> <during period="" starting="" the=""> <from 30="" days="" dose="" first="" last="" post="" to="" up="" vaccination=""> <after 30="" days="" dose="" end="" last="" post="" study="" to="" up="" vaccination=""><from end="" first="" study="" to="" vaccination=""><during entire="" period="" study="" the=""> (<total -="" 022="" cohort="" cohort,="" confirmed="" during="" episode="" hz="" total="" vaccinated="" zoster-006="">)</total></during></from></after></from></during></with></who></experiencing></with> | 29 |
| Template 23 | Number and percentage of subjects with <past><current> pre-<br/>existing medical conditions by SOC and PT (Total Vaccinated<br/>Cohort)</current></past> | 30 |
| Template 24 | Number and percentage of subjects who received study vaccine doses - by age sub-group (Total Vaccinated Cohort) | 30 |
| Template 25 | Number and percentage of subjects reporting the occurrence of<br><grade 3=""> <non-serious> <unsolicited adverse="" events=""> classified<br/>by MedDRA Primary System Organ Class and Preferred Term<br/><with causal="" relationship="" to="" vaccination=""> <with medically<br="">attended visit&gt; within the 30-day (Days 0-29) post-vaccination<br/>period - by age sub-group (<total cohort,="" total<br="" vaccinated="">Vaccinated Cohort - confirmed HZ episode during Zoster-<br/>006/022&gt;)</total></with></with></unsolicited></non-serious></grade> | 31 |
| Template 26 | Number and percentage of doses with <grade 3=""> unsolicited adverse events classified by MedDRA Primary System Organ</grade> | |

204486 (ZOSTER-056) Statistical Analysis Plan Final

| | Class and Preferred Term <with causal="" relationship="" to="" vaccination=""> <with attended="" medically="" visit=""> within the 30-day (Days 0-29) post-vaccination period - by age sub-group (Total Vaccinated Cohort)</with></with> | 31 |
|---|---|---|
| Template 27 | Global summary of <grade 3=""> <non-serious><unsolicited adverse="" events=""> <with causal="" relationship="" to="" vaccination=""> <with attended="" medically="" visit=""> reported <within (days="" 0-29)="" 30-day="" period="" post-vaccination="" the=""> - by age sub-group (Total Vaccinated Cohort)</within></with></with></unsolicited></non-serious></grade> | 32 |
| Template 28 | Number and percentage of subjects reporting the occurrence of <potential diseases="" immune-mediated=""> <serious adverse="" events=""> classified by MedDRA Primary System Organ Class <with causal="" relationship="" to="" vaccination=""> reported <from 30="" days="" dose="" first="" last="" post="" to="" up="" vaccination=""><after 30="" days="" dose="" end="" last="" post="" study="" to="" up="" vaccination=""> <from end="" first="" study="" until="" vaccination=""> - by age sub-group (<total -="" 022="" cohort="" cohort,="" confirmed="" during="" episode="" hz="" total="" vaccinated="" zoster-006="">)</total></from></after></from></with></serious></potential> | 32 |
| Template 29 | Number and percentage of subjects <with><experiencing> fatal SAEs classified by MedDRA Primary System Organ Class and Preferred Term <who died=""><with fatal="" of="" onset="" sae=""> <during period="" starting="" the=""> <from 30="" days="" dose="" first="" last="" post="" to="" up="" vaccination=""> <after 30="" days="" dose="" end="" last="" post="" study="" to="" up="" vaccination=""><from end="" first="" study="" the="" until="" vaccination=""><during entire="" period="" study="" the=""> by age sub-group (<total -="" 022="" cohort="" cohort,="" confirmed="" during="" episode="" hz="" total="" vaccinated="" zoster-006="">)</total></during></from></after></from></during></with></who></experiencing></with> | 33 |
| Template 30 | Number and percentage of subjects with <past><current> pre-<br/>existing medical conditions by SOC and PT – by age sub-group<br/>(Total Vaccinated Cohort)</current></past> | 34 |
| Template 31 | Listing of all SAEs from first vaccination until study end - by age sub-group (Total Vaccinated Cohort) | 34 |
| Template 32 | Listing of potential immune-mediated diseases (pIMDs) reported as identified by predefined list of preferred terms and/or by investigator assessment from first vaccination until study end - by age sub-group (Total Vaccinated Cohort) | 35 |
| Template 33 | Listing of dropouts due to AEs and SAEs from first vaccination until study end - by age sub-group (Total Vaccinated Cohort) | 35 |
| Template 34 | Listing of subjects who died during the entire study period – by age group (Total Enrolled Cohort) | 35 |
| Template 35 | Unsolicited adverse events classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period including number of events - SAE excluded (Total Vaccinated Cohort) | 36 |

204486 (ZOSTER-056) Statistical Analysis Plan Final

| Template 36 | Number (%) of subjects with serious adverse events from first vaccination until study end including number of events reported (Total Vaccinated Cohort) | 36 |
|---|---|---|
| Template 37 | Number and percentage of suspected HZ episodes (Total Vaccinated Cohort) | 36 |
| Template 38 | Number and percentage of suspected HZ episodes considering only subjects who had a confirmed HZ episode during Zoster-006/022 (Total Vaccinated Cohort) | 37 |
| Template 39 | Number and percentage of suspected HZ episodes - by age subgroup (Total Vaccinated Cohort) | 37 |
| Template 40 | Number and percentage of suspected HZ episodes considering only subjects who had a confirmed HZ episode during Zoster-006/022 - by age sub-group (Total Vaccinated Cohort) | 37 |
| Template 41 | Listing of subjects with a suspected HZ episode - by age subgroup (Total Vaccinated Cohort) | 38 |
| Template 42 | Listing of unsolicited adverse event within 30 days (Day 0-29) post receipt of only adjuvant - by age sub-group (Total Vaccinated Cohort) | 39 |

204486 (ZOSTER-056) Statistical Analysis Plan Final

#### **LIST OF ABBREVIATIONS**

AE Adverse event

CI Confidence Interval

CRF Case Report Form

CSR Clinical Study Report

CTRS Clinical Trial Registry Summary

HZ Herpes Zoster

LL Lower Limit of the confidence interval

MedDRA Medical Dictionary for Regulatory Activities

pIMD Potential Immune-Mediated Disease

SAE Serious adverse event

SAP Statistical Analysis Plan

SD Standard Deviation

Su Subunit

TFL Tables Figures and Listings

TOC Table of Content

TVC Total Vaccinated Cohort

UL Upper Limit of the confidence interval

YOA Years of age

#### 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|---|---|---|
| 26-FEB-2019 | Final version | Amendment 3 Final: |
| | Please note: As the SAP has been started long | 30-MAY-2017 |
| | back (19Dec2017) and reviewed also but was not | |
| | finalized due to study team change and delay in the | |
| | outcome of the Shingrix After Action Review (AAR) | |
| | post Type C meeting with CBER which was | |
| | required to be implemented in this SAP, the old | |
| | template of the SAP has been used. This has been | |
| | agreed by Lead Statistician. | |

#### 2. STUDY DESIGN

| One arm (HZ/su group), (n ~14,550) | | | | |
|---|---|---|---|---|
| Visit 1<br>Month 0<br>Vacc 1 | Visit 2<br>Month 2<br>Vacc 2 | Month 3<br>contact *<br>(SFU) | Month 8 Phone contact (SFU) | Month 14# Phone<br>contact<br>(SFU) |
| Follow-up period | | | | |

EPOCH 001

# i.e. 12 months post dose 2

n: number of subjects Vacc: vaccination SFU: Safety follow-up

- Experimental design: Phase IIIB open-label, non-randomised, multi-centric, multi-country cross-vaccination study, with a single group.
- Duration of the study: Approximately 14 months. Each subject will be followed for safety approximately 12 months after the second vaccine dose
  - Epoch 001: Primary starting at Visit 1 (Month 0) and ending at final phone contact (Month 14, i.e. 12 months post dose 2)
- Study groups:

Table 1 Study groups and epochs foreseen in the study

| Study Groups | Number of | Age (Min – Max) | Epochs |
|--------------|------------|------------------|-----------|
| Study Groups | subjects | Age (Will – Wax) | Epoch 001 |
| HZ/su Group | max 14,550 | > 50 YOA | Х |

<sup>\*</sup>Could be a visit or a phone contact.

Table 2 Study groups and treatment foreseen in the study

| Treatment name | Vaccine/Product name | Study Groups |
|----------------|----------------------|--------------|
| HZ/su | VZV gE | U7/au Craup |
| ΠZ/Su | AS01 <sub>B</sub> | HZ/su Group |

• Control: uncontrolled.

• Vaccination schedule: 0, 2 months.

• Treatment allocation: non-randomised.

• Blinding: open-label.

Table 3 Blinding of study epochs

| Study Epochs | Blinding |
|--------------|----------|
| Epoch 001 | open |

• Sampling schedule: no sampling.

• Type of study: self-contained.

• Data collection: electronic Case Report Form (eCRF).

#### 3. OBJECTIVES

#### 3.1. Primary objective

• To evaluate the safety, in terms of unsolicited Adverse Events (AEs), Serious Adverse Events (SAEs) and pIMD in all subjects, following administration of each dose of the HZ/su vaccine.

#### 3.2. Secondary objective

• To evaluate the incidence of suspected HZ episodes (self-reported or medically diagnosed) during the entire study period.

#### 4. ENDPOINTS

#### 4.1. Primary endpoints

- Occurrence of unsolicited AEs.
  - Occurrence, intensity and relationship to vaccination of unsolicited AEs during 30 days (Days 0-29) after each vaccination, according to the Medical Dictionary for Regulatory Activities (MedDRA) classification.
- Occurrence of SAEs.
  - Occurrence and relationship to vaccination of all SAEs from Month 0 until study end (Month 14, i.e. 12 months post dose 2).
- Occurrence of AEs of special interest.
  - Occurrence of any pIMDs from Month 0 until study end (Month 14, i.e. 12 months post dose 2).

#### 4.2. Secondary endpoints

- Occurrence of suspected HZ cases.
  - Occurrence of suspected HZ cases from Month 0 to study end.

#### 5. ANALYSIS SETS

#### 5.1. Definition

#### 5.1.1. Total Vaccinated Cohort

This study will collect only safety data. The statistical analysis of the safety endpoints will be based on the Total Vaccinated Cohort (TVC); hence no according to protocol (ATP) cohorts are defined for the purpose of statistical analysis.

The Total vaccinated cohort will include all subjects with at least one HZ/su vaccine administration documented for whom data are available:

• A safety analysis based on the Total vaccinated cohort will include all vaccinated subjects.

#### 5.2. Criteria for eliminating data from Analysis Sets

#### 5.2.1. Elimination from Total Vaccinated Cohort (TVC)

Code 900 (invalid informed consent or fraud data) and code 1030 (Study vaccine not administered at all) will be used for identifying subjects eliminated from Total Vaccinated Cohort.

#### 5.2.1.1. Excluded subjects

A subject will be excluded from the TVC analysis under the following conditions:

| Code | Condition under which the code is used |
|---|---|
| 900 | Invalid informed consent and fraud data |
| | (Subjects receiving a code 900 should not receive any other elimination codes) |
| 1030 | Study vaccine not administered at all |
| | (Subjects receiving a code 1030 should not receive any other elimination codes) |

#### 6. STATISTICAL ANALYSES

Note that standard data derivation rules and statistical methods are described in Section 11 and will not be repeated below.

#### 6.1. Demography

## 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

Demographic characteristics (age at first study vaccination in years, gender), withdrawal status will be summarised using descriptive statistics:

- Frequency tables will be generated for categorical variable such as centre.
- Mean, median, standard deviation will be provided for continuous data such as age, in Years, at vaccination in the current study.

#### 6.1.2. Additional considerations

- Demographic characteristics will also be tabulated by age sub-group at vaccination in the ZOSTER-056 (50-59, 60-69, 70-79 and ≥80 YOA).
- List of subjects withdrawn from vaccination with reason for withdrawal will be presented.
- The following table will be performed for web-disclosure:
  - Percentage of Enrolled subjects by country will be tabulated,
  - Percentage of Enrolled subjects in the following age categories ≤64, 65-84, ≥85 will be tabulated.

#### 6.2. Exposure

#### 6.2.1. Analysis of exposure planned in the protocol

Not applicable.

#### 6.2.2. Additional considerations

The number of doses administered will be tabulated overall and by age sub-group at vaccination in the ZOSTER-56 (50-59, 60-69, 70-79 and ≥80 YOA).

#### 6.3. Analysis of safety

#### 6.3.1. Analysis of safety planned in the protocol

The analysis for safety will be based on the TVC.

All analysis will be performed overall and by age sub-group at vaccination in the ZOSTER-056 (50-59, 60-69, 70-79 and  $\geq$ 80 YOA).

When appropriate, tabulations will be presented overall and by time of occurrence related to last vaccination (e.g. using windows such as Days 0-29 and more than 30 days post-vaccination

The results for the analysis of safety will be tabulated as follows:

- The proportion of subjects with at least one report of an unsolicited AE during the 30-day (Days 0–29) follow-up period after each vaccination classified according to the MedDRA System Organ Class and Preferred Terms will be tabulated, with exact 95% CI.
- The same tabulation will be performed for grade 3 unsolicited AEs (including SAEs) and for unsolicited AEs with a relationship to vaccination. The proportion of AEs resulting in a medically attended visit will also be tabulated.
- Total number/percentages of doses (per dose and overall) followed by AEs during the 30 days (Days 0-29) follow-up period after each vaccination classified according to the MedDRA System Organ Class and Preferred Terms will be tabulated.
- SAEs will be described in detail in listing for the entire study period.
- Withdrawal due to AE(s) and SAE will be described in detail in listing for the entire study period.
- Number of subjects with pIMDs will be tabulated according to the MedDRA System
  Organ Class and Preferred Terms for the period during first vaccination up to 30
  days post second vaccine dose, after 30 days post second vaccine dose to study end
  and from first vaccination to study end.

#### 6.3.2. Additional considerations

Following additional analyses will be performed:-

1. Number and percentage of subjects with at least one report of a grade 3 non-serious unsolicited AE during the 30-day (Days 0-29) follow-up period after each vaccination classified according to the MedDRA System Organ Class and Preferred Terms will be tabulated, with exact 95% CI.

- 2. Number and percentage of subjects reporting at least one SAE/ pIMD classified according to the MedDRA System Organ Class and Preferred Terms will be tabulated, with exact 95% CI with onset day of SAE during the time interval during study start to 30 days post 2<sup>nd</sup> vaccine dose, after 30 days post 2nd vaccine dose till study end and from study start till study end.
- 3. Number and percentage of subjects with fatal SAEs, classified by MedDRA Primary System Organ Class and Preferred Term will be presented with exact 95% CI in two ways:-
  - With onset of fatal SAE during the period starting from first vaccination to 30 days post last vaccination dose, after 30 days post last vaccination dose to study end and from first vaccination to study end
  - Who died during the period starting from first vaccination to 30 days post last vaccination dose, after 30 days post last vaccination dose to study end and entire study period.
- 4. Number and percentage of subjects reporting the occurrence of unsolicited adverse events classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period will also be presented, overall and by age sub-group with exact 95% CI on Total Vaccinated Cohort considering only subjects with a confirmed HZ episode during Zoster-006/022. The same tabulation will be performed for grade 3 unsolicited AEs and for unsolicited AEs with a relationship to vaccination.
- 5. Number and percentage of subjects reporting the occurrence of serious adverse event and pIMD, classified by MedDRA Primary System Organ Class and Preferred Term from first vaccination until study end will also be presented with exact 95% CI on Total Vaccinated Cohort considering only subjects with a confirmed HZ episode during Zoster-006/022.
- 6. List of subjects withdrawn from vaccination with reason for withdrawal will be presented from first vaccination until study end.
- 7. Listing of potential Immune-Mediated Diseases (pIMDs) reported as identified by predefined list of preferred terms and/or by investigator assessment from first vaccination until study end will be presented. Listing of the subjects who died will also be generated for the entire study period.
- 8. The unsolicited adverse events experienced within 30 days (Day 0-29) by subjects post receipt of only adjuvant will be presented in the listing.
- 9. Number and percentage of subjects with Past/Current pre-existing medical conditions by SOC and PT will be presented.

#### 6.4. Analysis of suspected HZ incidence

#### 6.4.1. Analysis of suspected HZ incidence planned in Protocol

1. The number of suspected HZ cases will be tabulated on TVC.

#### 6.4.2. Additional consideration

- 1. The analysis will also be performed on subjects having confirmed HZ episode from Zoster-006/022.
- 2. Listing for all the suspected HZ episodes will be presented.

#### 7. ANALYSIS INTERPRETATION

All analyses are descriptive.

#### 8. CONDUCT OF ANALYSES

#### 8.1. Sequence of analyses

| Description | Analysis<br>ID | Disclosure Purpose (CTRS=public posting, SR=study report, internal) | Dry run<br>review<br>needed<br>(Y/N) | Study Headline Summary (SHS)requiring expedited communication to upper management (Yes/No) | Reference for TFL |
|---|---|---|---|---|---|
| End of study | E1_01 | Study report | Y | Yes | Section 13 of the<br>SAP and TOC dated<br>26-FEB-19 |

#### 8.2. Statistical considerations for interim analyses

All analyses will be conducted on final data and therefore no statistical adjustment for interim analyses is required.

#### 9. CHANGES FROM PLANNED ANALYSES

Following are the changes from the planned analysis:-

- 1. As per protocol, it was mentioned that 'all analyses may be performed by age group at vaccination in the ZOSTER-006/022 (50-59, 60-69 and ≥70 YOA). However, team felt it is more reasonable to present the analysis based on age (by Year of birth) at first vaccination in current study. As the ≥ 80 YOA population in current study has increased in number because the cohort has aged, so the sub-group considered for the analysis has also been modified by dividing ≥70 YOA sub-group, further, into two (70-79 and ≥80 YOA) looking at the frequency of the subjects in these age groups (70-79 YOA = 3349 and ≥80 YOA = 2109). The age sub-group to be considered now will be (50-59, 60-69, 70-79 and ≥80 YOA)' based on the age (by Year of birth) at first vaccination in current study.
- 2. Table on presentation of fatal SAE has been added under additional consideration for safety analysis based on CBER feedback following Shingrix After Action Review (AAR) post Type C meeting with CBER.

- 3. Safety analysis by previous confirmed HZ episode (HZ episodes from Zoster-006/022 study) has been added.
- 4. Suspected HZ episodes in this study will also be presented on confirmed previous HZ episodes from Zoster-006/022 study.

## 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The TFL TOC provides the list of tables/listings and figures needed for the study report. It also identifies the tables eligible for the analysis and their role (synopsis, in-text, post-text, SHS, web disclosure). Note that all TFL aimed to be included as post-text are noted as post-text even if these are tabulation of individual data such as listing of SAE. The post-text material contains all source material for the study report and accordingly a post-text table may be redundant with an in-text table.

The following group name will be used in the TFLs:

| Group order in tables | Group label in tables | Group definition for footnote | Pooled Groups label in tables | Pooled definition for footnote |
|---|---|---|---|---|
| 1 | HZ/su | Herpes Zoster subunit vaccine | NA | NA |

NA=Not applicable

The following sub-group names will be used in the TFLs:

| Sub-group order in tables | Sub-group label in tables | Sub-group definition for footnote |
|---|---|---|
| 1 | 50-59YOA | Subjects aged 50-59 years* |
| 2 | 60-69YOA | Subjects aged 60-69 years* |
| 3 | 70-79YOA | Subjects aged 70-79 years |
| 4 | ≥80YOA | Subjects aged 80 years and over * |

<sup>\*</sup>age at first vaccination in Zoster-056 study

## 11. ANNEX 1 STANDARD DATA DERIVATION RULES AND STATISTICAL METHODS

#### 11.1. Statistical Method References

The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413].

#### 11.2. Standard data derivation

#### 11.2.1. Date derivation

- SAS date derived from a character date: In case day is missing, 15 is used. In case day and month are missing, 30 June is used.
- Onset day for an event (AE, medication, vaccination, ...): The onset day is the number of days between the last study vaccination and the onset/start date of the event. This is 0 for an event starting on the same day as a vaccination. See SAS date derived in case the start date of the event is incomplete.
- Duration: Duration of an event is expressed in days. It is the number of days between the start and the stop dates + 1. Therefore duration is 1 day for an event starting and ending on the same day.

#### 11.2.2. Dose number

- The study dose number is defined in reference to the number of study visits at which vaccination occurred. More specifically dose 1 refers to all vaccines administered at the first vaccination visit while dose 2 corresponds to all vaccinations administered at the second vaccination visit even if this is the first time a product is administered to the subject.
- Associated dose: the associated dose for an event (AE, medication,...) is the most recent study dose given before an event. In case the event takes place on the day a study dose is given, the associated dose will be that of the study dose, even if the event actually took place before vaccination. For instance, if an adverse event begins on the day of the study vaccination but prior to administration of the vaccine, it will be assigned to this dose. In case a study dose is not administered and an event occurs after the subsequent study dose (e.g. 2nd study dose), the associated dose of the event will be study dose associated to the subsequent study dose (e.g. dose 2).
- The number of doses for a product is the number of times the product was administered to a subject.
- The incidence per dose is the number of visits with vaccine administered at which an event was reported among all visits with vaccine administered.

#### 11.2.3. Demography

- For computation of age, following rule will be applied:-
  - Age will be calculated as the number of years between the date of birth and the date of first vaccination.
  - To ensure that the collection of date of birth will not jeopardise the privacy of Personally Identifiable Information (PII), only a partial date of birth (YYYY) will be collected. For calculation of age, as the date and month is not collected, the date will be replaced by the June 30th of the year. Accordingly, the age estimated using the middle of the year may differ by one year with the exact age.

#### 11.2.4. Safety

- For analysis of unsolicited adverse events, such as serious and non-serious adverse events by primary MedDRA term, and for the analysis of concomitant medications; all vaccinated subjects will be considered. Subjects who did not report any adverse event or any concomitant medication will be considered as subjects without an adverse event or concomitant medication respectively.
- HZ cases: Suspected HZ cases:
  - A <u>suspected HZ episode</u> is defined as a new rash characteristic of HZ (e.g., unilateral, dermatomal and accompanied by pain broadly defined to include allodynia, pruritus or other sensations).
  - Suspected HZ episode has to be confirmed by the investigator or the delegate judgement.

#### 11.3. Number of Decimals

The following decimal description from the decision rules will be used for the demography and safety analysis.

| Display Table | Parameters | Number of decimal digits |
|---|---|---|
| Demographic characteristics | Mean, median age | 1 |
| Demographic characteristics | SD (age) | 1 |
| All summaries | % of count, including LL & UL of CI | 1 |

#### 12. ANNEX 2: SUMMARY ON ELIMINATION CODES

Refer to section 5.

#### 13. ANNEX 3: STUDY SPECIFIC MOCK TFL

The following mock TFLs will be used.

The title and footnote are for illustration purpose and will be adapted to the study specificity as indicated in the TFL TOC.

Note that there may be few changes between the study specific SAP mock TFL and the final TFLs. These editorial/minor changes will not lead to a SAP amendment.

#### 13.1. Template of Tables and Figures

Template 1 Study population (Total Vaccinated Cohort)

| Number of subjects | HZ/su |
|---|---|
| Planned, N | |
| Vaccinated, N (Total Vaccinated Cohort) | |
| Completed, n (%) | |
| Demographics | HZ/su |
| N (Total Vaccinated Cohort) | |
| Females:Males | |
| Mean Age, years (SD) | |
| Median Age, years (minimum, maximum) | |
| <pre><most category="" frequent="" of="" race="">, n (%)</most></pre> | |
| <second category="" frequent="" most="" of="" race="">, n (%)</second> | |
| <third category="" frequent="" most="" of="" race="">, n (%)</third> | |

HZ/su = Herpes Zoster subunit vaccine

Completed = number of subjects who completed phone contact Month14

## Template 2 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Total Vaccinated Cohort)

| | ŀ | -lZ/su |
|-----------------------------------------------------------------|---|--------|
| | N | % |
| Number of subjects vaccinated | | |
| Number of subjects completed | | |
| Number of subjects withdrawn | | |
| Reasons for withdrawal : | | |
| Serious Adverse Event | | |
| Non-Serious Adverse Event | | |
| Protocol violation | | |
| Consent withdrawal (not due to an adverse event) | | |
| Migrated/moved from study area | | |
| Lost to follow-up (subjects with incomplete vaccination course) | | |
| Lost to follow-up (subjects with complete vaccination course) | | |
| Sponsor study termination | | |
| Suspected HZ episode | | |
| Others | | |

HZ/su = Herpes Zoster subunit vaccine

Vaccinated = number of subjects who were vaccinated in the study

Completed = number of subjects who completed last phone contact

Withdrawn = number of subjects who did not complete all visits up to last phone contact

n = number of subjects in a given category

% = (n / Number of subjects vaccinated) x 100

**Template 3** Summary of demographic characteristics (Total Vaccinated Cohort)

| | | HZ/su<br>N = | |
|---|---|---|---|
| Characteristics | Parameters or | Value or n | % |
| | Categories | | |
| Age (years) at vaccination dose : 1 | Mean | | |
| , | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| Gender | Female | | |
| | Male | | |
| Geographic Ancestry | African Heritage / African American | | |
| | American Indian or Alaskan Native | | |
| | Asian - Central/South Asian Heritage | | |
| | Asian - East Asian Heritage | | |
| | Asian - Japanese Heritage | | |
| | Asian - South East Asian Heritage | | |
| | Native Hawaiian or Other Pacific Islander | | |
| | White - Arabic / North African Heritage | | |
| | White - Caucasian / European Heritage | | |
| | Other | | |

HZ/su = Herpes Zoster subunit vaccine

N = total number of subjects

n/% = number / percentage of subjects in a given category

Value = value of the considered parameter

SD = standard deviation

#### Template 4 Number of subjects by center (Total Vaccinated Cohort)

| | | HZ/su | |
|-------------------------|---|-------|---|
| Center | N | | % |
| <each center=""></each> | | | |
| All | | | |

HZ/su = Herpes Zoster subunit vaccine

n = number of subjects for a given center or for all centers

All = sum of all subjects in total

 $% = n/AII \times 100$ 

Center = GSK Biologicals assigned center number

## Template 5 Number of subjects enrolled into the study as well as the number excluded from TVC analysis with reasons for exclusion

| | Total HZ/s | | <u>Z</u> /su | | | |
|---|---|---|---|---|---|---|
| Title | n | S | % | n | S | % |
| Total enrolled cohort | | | | | | |
| Invalid informed consent and fraud data (code 900) | | | | | | |
| Total effective cohort | | | | | | |
| Study vaccine dose not administrated but subject number allocated (code 1030) | | | | | | |
| Total vaccinated cohort | | | | | | |

HZ/su = Herpes Zoster subunit vaccine

Note: Subjects may have more than one elimination code assigned

n = number of subjects with the elimination code assigned excluding subjects who have been assigned a lower elimination code number

s = number of subjects with the elimination code assigned

% = percentage of subjects (n) relative to the Total vaccinated cohort

## Template 6 Number of subjects at each visit and list of withdrawn subjects (Total Vaccinated Cohort)

| Group | VISIT | N<br>(%) | Withdrawn<br>Subject numbers | Reason for withdrawal |
|---|---|---|---|---|
| HZ/su | VISIT 1 | | | |
| | VISIT 2 | | | |
| | VISIT 3 \ PHC M3 | | | |
| | PHONE CONT M8 | | | |
| | PHONE CONT M14 | | | |

HZ/su = Herpes Zoster subunit vaccine

N = Number of subjects who are still in the study up to the visit

Withdrawn = Subject who did not return after the visit

PHC = Phone contact

## Template 7 List of subjects withdrawn from vaccination with reason for withdrawal (Total Vaccinated Cohort)

| Group | Age | Subject number | Dose | Decision | Reason | Comment |
|-------|-----|----------------|------|----------|--------|---------|
| HZ/su | | | | | | |

HZ/su = Herpes Zoster subunit vaccine

## Template 8 Deviations from specifications for intervals between study visits (Total Vaccinated Cohort)

| | | VISIT 1 – VISIT 2 | VISIT 2 - VISIT 3\PHC | VISIT 2 – PHONE | VISIT 2 – PHONE CONT |
|---|---|---|---|---|---|
| | | | M3 | CONT M8 | M14 |
| Group | | Protocol | Protocol | Protocol | Protocol |
| | | from 49 to 83<br>days | from 30 to 48 days | from 180 to 240 days | from 335 to 395 days |
| HZ/su | N | | | | |
| | n | | | | |
| | % | | | | |
| | range | _ | | | |

HZ/su = Herpes Zoster subunit vaccine

N = total number of subjects with available results

n/% = number / percentage of subjects with results outside of the interval

range = minimum-maximum for intervals

PHC = Phone contact

#### Template 9 Number of enrolled subjects by country

| | | HZ/su<br>N = |
|-----------------|--------------------------|--------------|
| Characteristics | Categories | n |
| Country | <each country=""></each> | |

HZ/su = Herpes Zoster subunit vaccine

N = Number of enrolled subjects

n= number of enrolled subjects for a given country or for all countries

#### Template 10 Number of enrolled subjects by age category

| | | HZ/su<br>N = |
|-----------------|----------------------|--------------|
| Characteristics | Categories | N |
| Age category | Adults (18-64 years) | |
| | From 65-84 years | |
| | 85 years and over | |
| | Missing | |

HZ/su = Herpes Zoster subunit vaccine

N = Number of enrolled subjects

n= number of enrolled subjects included for a given age category or for all age categories Missing = Subjects enrolled in the study but did not receive the first vaccine dose at Month 0

Template 11 Minimum and maximum activity dates (Total Vaccinated Cohort)

| Group | Activity number | Activity Description | Minimum date | Maximum date |
|-------|-----------------|----------------------|--------------|--------------|
| HZ/su | 110 | VISIT 1 | | |
| | 120 | VISIT 2 | | |
| | 210 | VISIT 3 \ PHC M3 | | |
| | 220 | PHONE CONT M8 | | |
| | 230 | PHONE CONT M14 | | |

HZ/su = Herpes Zoster subunit vaccine

PHC = Phone contact

204486 (ZOSTER-056) Statistical Analysis Plan Final

#### Template 12 Study population – by age sub-group (Total Vaccinated Cohort)

| [each age sub-group] |
|----------------------|
| - |
| [each age sub-group] |

Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80 years and over

HZ/su = Herpes Zoster subunit vaccine

Completed = number of subjects who completed last phone contact

Template 13 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal – by age sub-group (Total Vaccinated Cohort)

| | [each a | ge sub-group] | Total | |
|---|---|---|---|---|
| | n | % | n | % |
| Number of subjects vaccinated | | | | |
| Number of subjects completed | | | | |
| Number of subjects withdrawn | | | | |
| Reasons for withdrawal : | | | | |
| Serious Adverse Event | | | | |
| Non-Serious Adverse Event | | | | |
| Protocol violation | | | | |
| Consent withdrawal (not due to an adverse event) | | | | |
| Migrated/moved from study area | | | | |
| Lost to follow-up (subjects with incomplete vaccination course) | | | | |
| Lost to follow-up (subjects with complete vaccination course) | | | | |
| Sponsor study termination | | | | |
| Suspected HZ episode | | | | |
| Others | | | | |

<sup>\*</sup>Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80 years and over

HZ/su = Herpes Zoster subunit vaccine

Vaccinated = number of subjects who were vaccinated in the study

Completed = number of subjects who completed last phone contact

Withdrawn = number of subjects who did not complete all visits up to last phone contact

n = number of subjects in a given category

% = (n / Number of subjects vaccinated) x 100

## Template 14 Summary of demographic characteristics - by age sub-group (Total Vaccinated Cohort)

| | | [each age sub-<br>group]<br>N = | | Total<br>N = | |
|---|---|---|---|---|---|
| Characteristics | Parameters or | Value or | % | Value or n | % |
| | Categories | n | | | |
| Age (years) at vaccination dose: 1 | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Minimum | | | | |
| | Maximum | | | | |
| Gender | Female | | | | |
| | Male | | | | |
| Geographic Ancestry | African Heritage / African American | | | | |
| | American Indian or Alaskan Native | | | | |
| | Asian - Central/South Asian Heritage | | | | |
| | Asian - East Asian Heritage | | | | |
| | Asian - Japanese Heritage | | | | |
| | Asian - South East Asian Heritage | | | | |
| | Native Hawaiian or Other Pacific Islander | | | | |
| | White - Arabic / North African Heritage | | | | |
| | White - Caucasian / European Heritage | | | | |
| | Other | | | | |

<sup>\*</sup>Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80 years and over

HZ/su = Herpes Zoster subunit vaccine

N = total number of subjects

n/% = number / percentage of subjects in a given category

Value = value of the considered parameter

SD = standard deviation

Note that the exact age is unknown since only the year of date of birth is recorded. Accordingly, the age estimated using the middle of the year may differ by one year with the exact age

Template 15 Number of subjects by center - by age sub-group (Total Vaccinated Cohort)

| | [each subgroup] | | Total |
|-------------------------|-----------------|---|-------|
| Center | N | N | % |
| <each center=""></each> | | | |
| All | | | |

\*Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80 years and over

HZ/su = Herpes Zoster subunit vaccine

n = number of subjects for a given center or for all centers

All = sum of all subjects in total

 $% = n/AII \times 100$ 

Center = GSK Biologicals assigned center number

## Template 16 Number of subjects at each visit and list of withdrawn subjects by - age sub-group (Total Vaccinated Cohort)

| [each age<br>sub-<br>group] | Group | VISIT | Withdrawn<br>Subject numbers | Reason for withdrawal |
|---|---|---|---|---|
| | HZ/su | VISIT 1 | | |
| | | VISIT 2 | | |
| | | VISIT 3 \ PHC M3 | | |
| | | PHONE CONT M8 | | |
| | | PHONE CONT M14 | | |

\*Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80 years and over

HZ/su = Herpes Zoster subunit vaccine

N = Number of subjects who are still in the study up to the visit

Withdrawn = Subject who did not return after the visit

PHC = Phone contact

Template 17 Number and percentage of subjects who received study vaccine doses (Total Vaccinated Cohort)

| | HZ/su<br>N = | |
|--------------------------------|--------------|---|
| Total number of doses received | N | % |
| 1 | | |
| 2 | | |
| Any | | |

HZ/su = Herpes Zoster subunit vaccine

N = number of subjects in the group or in total included in the considered cohort

n/% = number/percentage of subjects receiving the specified total number of doses

Any = number and percentage of subjects receiving at least one dose

Template 18 Number and percentage of subjects reporting the occurrence of <grade 3> <non-serious><unsolicited adverse events> classified by MedDRA Primary System Organ Class and Preferred Term <with causal relationship to vaccination> <with medically attended visit> within the 30-day (Days 0-29) post-vaccination period (<Total Vaccinated Cohort, Total Vaccinated Cohort - confirmed HZ episode during Zoster-006/022>)

| | | | | Z/su<br>1 = | |
|---|---|---|---|---|---|
| | | | | 959 | % CI |
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n | % | LL | UL |
| At least one symptom | | | | | |
| Each SOC | At least one PT related to the corresponding SOC | | | | |
| | Each PT | | | | |

HZ/su = Herpes Zoster subunit vaccine

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n/%= number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

204486 (ZOSTER-056) Statistical Analysis Plan Final

Template 19 Number and percentage of doses with <grade 3> unsolicited adverse events classified by MedDRA Primary System Organ Class and Preferred Term <with causal relationship to vaccination> <with medically attended visit> within the 30-day (Days 0-29) post-vaccination period (Total Vaccinated Cohort)

| | | | HZ/s | | |
|---|---|---|---|---|---|
| | | 95% | | 6 CI | |
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n | % | LL | UL |
| At least one symptom | | | | | |
| Each SOC | At least one PT related to the corresponding SOC | | | | |
| | Each PT | | | | |

HZ/su = Herpes Zoster subunit vaccine

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of administered doses

n/% = number/percentage of doses with the symptom

95% CI= exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Template 20 Global summary of <grade 3> <non-serious><unsolicited adverse events> <with causal relationship to vaccination> <with medically attended visit> reported within the 30-day (Days 0-29) post-vaccination period (Total Vaccinated Cohort)

| | HZ/su |
|---------------------------------------------------------------------|-------|
| Number of subjects with at least one unsolicited symptom reported | |
| Number of doses followed by at least one unsolicited symptom | |
| Number of unsolicited symptoms classified by MedDRA Preferred Term* | |
| Number of unsolicited symptoms reported** | |

HZ/su = Herpes Zoster subunit vaccine

<sup>\*</sup> Symptoms reported by a subject after a given dose and classified by the same Preferred Term are counted once

<sup>\*\*</sup> Symptoms reported by a subject after a given dose and classified by the same Preferred Term and the same start date of the event, are counted once

Template 21 Number and percentage of subjects reporting the occurrence of <potential Immune-Mediated Diseases> <serious adverse events> classified by MedDRA Primary System Organ Class and Preferred Term <with causal relationship to vaccination> reported <from first vaccination up to 30 days post last vaccination dose> <after 30 days post last vaccination dose up to study end> <from first vaccination until study end > (<Total Vaccinated Cohort, Total Vaccinated Cohort - confirmed HZ episode during Zoster-006/022>)

| | | HZ/su<br>N = | | | | |
|---|---|---|---|---|---|---|
| | | | | | 95% | <b>6 CI</b> |
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n* | n | % | LL | UL |
| At least one symptom | | | | | | |
| Each SOC | At least one PT related to the corresponding SOC Each PT | | | | | |

HZ/su = Herpes Zoster subunit vaccine group

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n/%= number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

n\* = number of events reported (only required for CTRS posting)

Template 22 Number and percentage of subjects <with><experiencing> fatal SAEs classified by MedDRA Primary System Organ Class and Preferred Term <who died> <with onset of fatal SAE> <during the period starting> <from first vaccination up to 30 days post last vaccination dose> <after 30 days post last vaccination dose up to study end> <from first vaccination to study end > <during the entire study period> (<Total Vaccinated Cohort, Total Vaccinated Cohort - confirmed HZ episode during Zoster-006/022>)

| | | | HZ<br>N | /su<br>= | |
|---|---|---|---|---|---|
| | | ! | | 95% | 6 CI |
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n | % | LL | UL |
| At least one symptom | | | | | |
| Each SOC | At least one PT related to the corresponding SOC | | | | |
| | Each PT | | | | |

HZ/su = Herpes Zoster subunit vaccine

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n/%= number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

#### Template 23 Number and percentage of subjects with <past><current> preexisting medical conditions by SOC and PT (Total Vaccinated Cohort)

| | | Н | |
|---|---|---|---|
| SOC (CODE) | PT (CODE) | n | % |
| At least one condition | | | |
| Blood and lymphatic system disorders (10005329) | Any condition | | |
| | Anaemia (10002034) | | |
| Cardiac disorders (10007541) | Any condition | | |
| , , | Angina pectoris (10002383) | | |
| | Arrhythmia (10003119) | | |
| | Atrial fibrillation (10003658) | | |
| | Cardiac failure (10007554) | | |
| | Coronary artery disease (10011078) | | |
| | Hypertensive heart disease (10020823) | | |
| | Myocardial ischaemia (10028600) | | |
| Each SOC (CODE) | Any condition | | |
| | Each PT (CODE) | | |

HZ/su = Herpes Zoster subunit vaccine

N = total number of subjects

n/% = number / percentage of subjects reporting the condition at least once

Template 24 Number and percentage of subjects who received study vaccine doses - by age sub-group (Total Vaccinated Cohort)

| | [each age sub-group]* | | | Total |
|--------------------------------|-----------------------|---|---|-------|
| Total number of doses received | N | % | N | % |
| 1 | | | | |
| 2 | | | | |
| Any | | | | |

\*Age sub-group is based on subject's age at first dose of vaccination in Zoster-056

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80 years and over

HZ/su = Herpes Zoster subunit vaccine

N = number of subjects in each sub-group or in total included in the considered cohort

n/% = number/percentage of subjects receiving the specified total number of doses

Any = number and percentage of subjects receiving at least one dose

Template 25 Number and percentage of subjects reporting the occurrence of <grade 3> <non-serious> <unsolicited adverse events> classified by MedDRA Primary System Organ Class and Preferred Term <with causal relationship to vaccination> <with medically attended visit> within the 30-day (Days 0-29) post-vaccination period - by age subgroup (<Total Vaccinated Cohort, Total Vaccinated Cohort - confirmed HZ episode during Zoster-006/022>)

| | | [ea | ch age s<br>HZ/s<br>N : | su | nb] |
|---|---|---|---|---|---|
| | | 95 | | 95% | 6 CI |
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n | % | LL | UL |
| At least one symptom | | | | | |
| Each SOC | At least one PT related to the corresponding SOC | | | | |
| | Each PT | | | | |

<sup>\*</sup>Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80 years and over

HZ/su = Herpes Zoster subunit vaccine

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n/%= number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Template 26 Number and percentage of doses with <grade 3> unsolicited adverse events classified by MedDRA Primary System Organ Class and Preferred Term <with causal relationship to vaccination> <with medically attended visit> within the 30-day (Days 0-29) post-vaccination period - by age sub-group (Total Vaccinated Cohort)

| | | [eacl | [each age sub-group] | | |
|---|---|---|---|---|---|
| | | | HZ/su | | |
| | | | N = | | |
| | | 95 | | 95% | % CI |
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n | % | LL | UL |
| At least one symptom | | | | | |
| Each SOC | At least one PT related to the corresponding | | | | |
| | SOC | | | | |
| | Each PT | | | | |

<sup>\*</sup>Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80 years and over

HZ/su = Herpes Zoster subunit vaccine

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of administered doses

n/% = number/percentage of doses with the symptom

95% CI= exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Template 27 Global summary of <grade 3> <non-serious><unsolicited adverse events> <with causal relationship to vaccination> <with medically attended visit> reported <within the 30-day (Days 0-29) post-vaccination period> - by age sub-group (Total Vaccinated Cohort)

| | [each age sub-<br>group]* | All |
|---|---|---|
| Number of subjects with at least one unsolicited symptom reported | | |
| Number of doses followed by at least one unsolicited symptom | | |
| Number of unsolicited symptoms classified by MedDRA Preferred Term* | | |
| Number of unsolicited symptoms reported** | | |

<sup>\*</sup>Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80 years and over

HZ/su = Herpes Zoster subunit vaccine

Template 28 Number and percentage of subjects reporting the occurrence of <potential Immune-Mediated Diseases> <serious adverse events> classified by MedDRA Primary System Organ Class <with causal relationship to vaccination> reported <from first vaccination up to 30 days post last vaccination dose vafter 30 days post last vaccination dose up to study end> <from first vaccination until study end> - by age sub-group (<Total Vaccinated Cohort, Total Vaccinated Cohort - confirmed HZ episode during Zoster-006/022>)

| | | [eac | h age sul<br>N= | o-grou | ıp]* |
|---|---|---|---|---|---|
| | | | | 95% | % CI |
| Primary System Organ Class (CODE) | Preferred Term (CODE) | N | % | LL | UL |
| At least one symptom | | | | | |
| Each SOC | At least one PT related to the corresponding | | | | |
| | SOC | | | | |
| | Each PT | | | | |

<sup>\*</sup>Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80 years and over

HZ/su = Herpes Zoster subunit vaccine

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n/%= number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

<sup>\*</sup> Symptoms reported by a subject after a given dose and classified by the same Preferred Term are counted once

<sup>\*\*</sup> Symptoms reported by a subject after a given dose and classified by the same Preferred Term and the same start date of the event, are counted once

Template 29 Number and percentage of subjects <with><experiencing> fatal SAEs classified by MedDRA Primary System Organ Class and Preferred Term <who died><with onset of fatal SAE> <during the period starting> <from first vaccination up to 30 days post last vaccination dose > <after 30 days post last vaccination dose up to study end><from first vaccination until the study end><during the entire study period> by age sub-group (<Total Vaccinated Cohort, Total Vaccinated Cohort - confirmed HZ episode during Zoster-006/022>)

| | | [eac | h age su<br>N= | | 1b]* |
|---|---|---|---|---|---|
| | | 959 | | % CI | |
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n | % | LL | UL |
| At least one symptom | | | | | |
| Each SOC | At least one PT related to the corresponding SOC | | | | |
| | Each PT | | | | |

\*Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80 years and over

HZ/su = Herpes Zoster subunit vaccine

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n/%= number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Please note this table will be generated only based on final feedback and agreement with CBER

#### Template 30 Number and percentage of subjects with <past><current> preexisting medical conditions by SOC and PT – by age sub-group (Total Vaccinated Cohort)

| | | | [each age sub-<br>group]*<br>N= | | Total<br>N= |
|---|---|---|---|---|---|
| SOC (CODE) | PT (CODE) | N | % | N | % |
| At least one condition | | | | | |
| Blood and lymphatic system disorders (10005329) | Any condition | | | | |
| , | Anaemia (10002034) | | | | |
| Cardiac disorders (10007541) | Any condition | | | | |
| | Angina pectoris (10002383) | | | | |
| | Arrhythmia (10003119) | | | | |
| | Atrial fibrillation (10003658) | | | | |
| | Cardiac failure (10007554) | | | | |
| | Coronary artery disease (10011078) | | | | |
| | Hypertensive heart disease (10020823) | | | | |
| | Myocardial ischaemia (10028600) | | | | |
| Each SOC (CODE) | Any condition | | | | |
| | Each PT (CODE) | | | | |

<sup>\*</sup>Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80 years and over

HZ/su = Herpes Zoster subunit vaccine group

N = total number of subjects

n/% = number / percentage of subjects reporting the condition at least once

Template 31 Listing of all SAEs from first vaccination until study end - by age sub-group (Total Vaccinated Cohort)

| Goup | Sub-<br>group<br>* | Sub.No | Age<br>at<br>onse<br>t<br>(Year | Se<br>x | Verbati<br>m | Preferre<br>d term | Syste<br>m<br>Organ<br>Class | D | е | Day<br>of<br>onse<br>t | Duratio<br>n | Intensit<br>y | Causalit<br>y | Outcom<br>e |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| [HZ/s<br>u | [each<br>age<br>sub-<br>group] | | · | | | | | | | | | | | |

<sup>\*</sup>Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80 years and over

HZ/su = Herpes Zoster subunit vaccine group

MED = Medically attended visit

HO = Hospitalization,

MD = medical personnel

Please note this listing will also include the SAE related to only adjuvants which subject has received

# Template 32 Listing of potential immune-mediated diseases (pIMDs) reported as identified by predefined list of preferred terms and/or by investigator assessment from first vaccination until study end - by age subgroup (Total Vaccinated Cohort)

| Group | Sub-group | Patient ID | Country | Age at onset (Y) | Gender | Primary System<br>Organ Class | Preferred term |
|---|---|---|---|---|---|---|---|
| HZ/su | [each age | | | | | | |
| | sub-group] | | | | | | |

| Group | Sub-group* | Dose | Day of onset | Serious pIMD based on Investigator? | SAE<br>(Y/N) | Outcome | pIMD<br>Source |
|---|---|---|---|---|---|---|---|
| HZ/su | [each age | | | | | | |
| | sub-group] | | | | | | |

<sup>\*</sup>Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80 years and over

HZ/su = Herpes Zoster subunit vaccine

Template 33 Listing of dropouts due to AEs and SAEs from first vaccination until study end - by age sub-group (Total Vaccinated Cohort)

| Group | Sub- | Study- | Country | Gender | Race | AE | SAE | Causality | Outcome | Type of |
|---|---|---|---|---|---|---|---|---|---|---|
| | group* | Subject | | | | Description | | | | discontinuation |
| | | No. | | | | | | | | |
| HZ/su | [each age | | | | | | | | | |
| | sub-group] | | | | | | | | | |

<sup>\*</sup>Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80 years and over

HZ/su = Herpes Zoster subunit vaccine

Type of discontinuation = discontinuation from study or from treatment

Template 34 Listing of subjects who died during the entire study period – by age group (Total Enrolled Cohort)

| Grou | Sub | Se | Countr | Rac | Age | Verbati | Preferre | Primar | ME | Dos | Days | Dos | Days | SAE | SAE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| p | | X | у | е | at | m | d term | , | | | | | | | Causalit |
| | No. | | | | Onse<br>t<br>(Year<br>) | | | - | e | to<br>onse<br>t of<br>fatal | of fatal<br>SAE | to<br>deat<br>h | n death<br>and<br>previou<br>s dose | n | У |
| HZ/su | X1 | | | | | | | | НО | | | | | | |
| | X2 | | | | | | | | НО | | | | | | |
| | X3 | | | | | | | | НО | | | | | | |

HZ/su = Herpes Zoster subunit vaccine

No Group= Enrolled not vaccinated

MED = Medical Advice type (HO: hospitalisation, ER: emergency room visit, MD: medical practice visit)

# Template 35 Unsolicited adverse events classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period including number of events - SAE excluded (Total Vaccinated Cohort)

| | | | HZ/s<br>N = | |
|---|---|---|---|---|
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n* | N | % |
| At least one symptom | | | | |
| <each soc=""></each> | <each pt="" term=""></each> | | | |

HZ/su = Herpes Zoster subunit vaccine

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with at least one administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

Template 36 Number (%) of subjects with serious adverse events from first vaccination until study end including number of events reported (Total Vaccinated Cohort)

| | | | HZ/su<br>N = | | |
|---|---|---|---|---|---|
| Type of Event | Primary System Organ Class | Preferred Term (CODE) | n* | N | % |
| SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Related SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Fatal SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Related fatal SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |

HZ/su = Herpes Zoster subunit vaccine group

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the event at least once

Template 37 Number and percentage of suspected HZ episodes (Total Vaccinated Cohort)

| | | HZ/su<br>N = |
|---------------------------|---|--------------|
| Categories | n | % |
| HZ episode | | |
| Suspected HZ episode only | | |
| Confirmed HZ episode | | |

HZ/su = Herpes Zoster subunit vaccine

N = total number of subjects

n/% = number / percentage of subjects in a given category

HZ episode: number of subjects with at least one suspected episode

Suspected HZ episode only: Suspected HZ episode not confirmed by the Investigator/Delegate

Confirmed HZ episode: Suspected HZ episode confirmed by the Investigator/Delegate

## Template 38 Number and percentage of suspected HZ episodes considering only subjects who had a confirmed HZ episode during Zoster-006/022 (Total Vaccinated Cohort)

| | | HZ/su<br>N = |
|---------------------------|---|--------------|
| Categories | n | % |
| HZ episode | | |
| Suspected HZ episode only | | |
| Confirmed HZ episode | | |

HZ/su = Herpes Zoster subunit vaccine

N = total number of placebo subjects from Zoster-006/022 (TVC) with a confirmed HZ episode during Zoster-006/022 vaccinated in this study

n/% = number / percentage of subjects in a given category

HZ episode: number of subjects with at least one suspected episode

Suspected HZ episode only: Suspected HZ episode not confirmed by the Investigator/Delegate

Confirmed HZ episode: Suspected HZ episode confirmed by the Investigator/Delegate

Template 39 Number and percentage of suspected HZ episodes - by age subgroup (Total Vaccinated Cohort)

| | [each age sub-<br>group]*<br>N= | | | otal<br> = |
|---|---|---|---|---|
| Categories | n | % | N | % |
| HZ episode | | | | |
| Suspected HZ episode only | | | | |
| Confirmed HZ episode | | | | |

\*Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80years and over

HZ/su = Herpes Zoster subunit vaccine

N = total number of subjects

n/% = number / percentage of subjects in a given category

HZ episode: number of subjects with at least one suspected episode

Suspected HZ episode only: Suspected HZ episode not confirmed by the Investigator/Delegate

Confirmed HZ episode: Suspected HZ episode confirmed by the Investigator/Delegate

Template 40 Number and percentage of suspected HZ episodes considering only subjects who had a confirmed HZ episode during Zoster-006/022 - by age sub-group (Total Vaccinated Cohort)

| | [each age sub-<br>group]*<br>N= | | Total<br>N= |
|---|---|---|---|
| Categories | n % | N | % |
| HZ episode | | | |
| Suspected HZ episode only | | | |
| Confirmed HZ episode | | | |

\*Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80years and over

HZ/su = Herpes Zoster subunit vaccine

204486 (ZOSTER-056) Statistical Analysis Plan Final

N = total number of placebo subjects from Zoster-006/022 (TVC) with a confirmed HZ episode during Zoster-006/022 and vaccinated in this study

n/% = number / percentage of subjects in a given category

HZ episode: number of subjects with at least one suspected episode

Suspected HZ episode only: Suspected HZ episode not confirmed by the Investigator/Delegate

Confirmed HZ episode: Suspected HZ episode confirmed by the Investigator/Delegate

## Template 41 Listing of subjects with a suspected HZ episode - by age sub-group (Total Vaccinated Cohort)

| Grou<br>p | Sub-<br>group* | Patient<br>ID | Countr<br>y | vaccination in | HZ<br>episode<br>number | Rash<br>start<br>date | Start date of pain/itching/abnor mal sensation at rash site |
|---|---|---|---|---|---|---|---|
| HZ/su | [each | | | | | | |
| | age sub- | | | | | | |
| | group] | | | | | | |

| Grou<br>p | Sub-<br>grou<br>p | Confirme<br>d by<br>INV/DEL | first<br>vaccinatio<br>n in | Date of<br>second<br>vaccinatio<br>n in<br>Zoster-056 | s dose | h | End date of pain/itching/abnorm al sensation at rash site |
|---|---|---|---|---|---|---|---|
| | [each<br>age<br>sub-<br>group<br>] | | | | | | |

<sup>\*</sup>Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80 years and over

HZ/su = Herpes Zoster subunit vaccine

INV/DEL = Investigator/Delegate

HZ\_P30D2 = flag for suspected HZ episode occurring after 30 days post-Dose 2

204486 (ZOSTER-056) Statistical Analysis Plan Final

## Template 42 Listing of unsolicited adverse event within 30 days (Day 0-29) post receipt of only adjuvant - by age sub-group (Total Vaccinated Cohort)

| Goup St | roup | Age<br>at<br>onset<br>(Year | X | Verbati<br>m | Preferre<br>d term | Syste<br>m<br>Organ<br>Class | ME<br>D<br>type | е | Day<br>of<br>onse | Duratio<br>n | Intensit<br>y | Causalit<br>y | Outcom<br>e |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| u ag | each<br>ge<br>ub-<br>roup] | | | | | | | | | | | | |

\*Age sub-group is based on subject's age at first vaccination

50-59YOA = Subjects aged 50-59 years

60-69YOA = Subjects aged 60-69 years

70-79YOA = Subjects aged 70-79 years

≥80YOA = Subjects aged 80 years and over

HZ/su = Herpes Zoster subunit vaccine group

MED = Medically attended visit

HO = Hospitalization,

MD = medical personnel